CLINICAL TRIAL: NCT05637073
Title: Impact of the Type of Treatment of the Endometrioma on Ovarian Reserve
Brief Title: Effect of Management of the Endometrioma on Ovarian Reserve
Acronym: IMTERO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Collaborators: Hospital Comarcal Francesc de Borja Gandía, Valencia, Spain (Unknown); Hospital Universitario San Juan de Alicante (Other); Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Antonio Cano Sanchez, Professor Obstetrics & Gynecology, University of Valencia
Other Study IDs: IMTERO_22
Record Dates: First submitted 2022-10-22; First posted 2022-12-05 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Endometrioma
MeSH Terms: conditions — Endometriosis | interventions — dienogest; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Serum will be stored for measurement of AMH levels in a central laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Dienogest — Some women in the cohort will be treated with dienogest for one year after consensus with the physician
Procedure: Laparoscopic cystectomy — Some women in the cohort will be treated with laparoscopic cystectomy after consensus with the physician
Other: Control with ultrasound without other type of intervention — Some women in the cohort will be followed with ultrasound control, without other intervention, after consensus with the physician

SUMMARY:
Investigators aimed at comparing the impact on ovarian reserve of three usual-care management options of endometrioma, laparoscopic cystectomy (LC), hormonal treatment with daily dienogest (HT), or mere ultrasound control (UC).

Ovarian reserve will be measured by the effect on the circulating levels of anti-Mullerian hormone (AMH). Secondary objectives will be effect on pelvic pain, other symptoms, sexual function, quality of life, progression in size of the endometrioma, impact on work productivity and activity impairment, and satisfaction with treatment.

Participants will be followed by up to one year.

DETAILED DESCRIPTION:
Investigators aimed at comparing the impact on ovarian reserve of three usual-care management options of endometrioma, laparoscopic cystectomy (LC), hormonal treatment with daily dienogest (HT), or mere ultrasound control (UC).

Secondary objectives were the comparison of the effect on i) pelvic pain, including dysmenorrhea, non-menstrual pelvic pain, deep dyspareunia, or dyschezia, ii) other symptoms including menorrhagia, gastrointestinal symptoms different to dyschezia, or urinary symptoms; iii) quality of life as assessed by the EHP-30 questionnaire; iv) sexual functions, as assessed the female sexual function index (FSFI); v) progression in the size of the tumor in the case of the two non-surgical approaches; vi) impact on work productivity and activity impairment; vii) satisfaction in the patient.

A prospective assessment will be performed on a cohort of women with endometrioma diagnosed by ultrasound from diagnosis for up to one year. The assignment to each management option will be performed under usual care conditions so that the selected option will result from the shared clinical decision of the clinician with the patient.

The target population will be composed of Caucasian premenopausal women between 18-39 years with the diagnosis of endometrioma, one or more, with a diameter of up to 7 cm by endovaginal ultrasound. Body mass index comprised between 17-30 Kg/m2.

Participants will be controlled at 3 months, 6 months and one year.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian premenopausal women between 18-39 years with the diagnosis of endometrioma, one or more, with a diameter of up to 7 cm by endovaginal ultrasound. Body mass index comprised between 17-30 Kg/m2

Exclusion Criteria:

* Previous ovarian surgery;
* Previous pathologies involving the ovary, including other ovarian tumors, polycystic ovaries, or pelvic inflammatory disease;
* Previous diagnosis of cancer treated with chemotherapy or local radiotherapy;
* Diseases affecting the endocrine system, diabetes, thyroid, hyperprolactinemia, or the immune system (lupus, Crohn,…);
* Genesic wish;
* Endometrioma >7 cm;
* Unhealthy habits, including smoking, alcohol consumption above social level, or illicit drugs;
* Insufficient level of autonomy for unrestrictedly signing informed consent;
* Current or previous use of hormonal contraceptives, Gonadotropin-Releasing Hormone (GnRH) analogues, any drug with a known effect on endometriosis, or any drug under investigation, for what a washing up period of 6 months will be required in all cases.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Caucasian premenopausal women between 18-39 years with the diagnosis of endometrioma, one or more, with a diameter of up to 7 cm by endovaginal ultrasound. Body mass index comprised between 17-30 Kg/m2.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-11-02 (Estimated); Study Completion 2024-11-02 (Estimated)

PRIMARY OUTCOMES:
Change in the levels of anti-Mullerian hormone | Change from baseline AMH levels at 1 year
  Ovarian reserve as measured by the levels of AMH

SECONDARY OUTCOMES:
Change of Pelvic pain | Change from baseline pelvic pain at 1 year.
  Dysmenorrhea, non-menstrual pelvic pain, deep dyspareunia, or dyschezia measured by a visual analogue scale from 0 to 5 and in which higher score means worse outcome.
Change in quality of life | Change from baseline EHP-30 score at 1 year.
  Assessed by the Endometriosis Health Profile-30 (EHP-30) questionnaire, in which the minimum score is 0 and the highest 150. Higher score means a worse outcome.
Change in sexual function | Change from baseline FSFI score at 1 year.
  Assessed the female sexual function index (FSFI) questionnaire in which there are 6 questions from 0 to 5. The highest score is 30 and the lowest 0. Lower score means worse outcome.
Change in volume of the tumor | Change from baseline endometrioma volume at 1 year.
  Measured by ultrasound, in the case of the two non-surgical approaches
Satisfaction of the patient | Satisfaction level measured by Likert scale at 1 year.
  Satisfaction as assessed by a Likert scale in which the score is from 0 to 5 in which higher score means better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital Poznan, Poznan, Poland
- Hosp Clinico Universitario-INCLIVA, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided